CLINICAL TRIAL: NCT06489106
Title: Optimization of Noninvasive Spinal Stimulation to Restore Hand Function in Children with Spinal Cord Injury
Brief Title: Noninvasive Spinal Stimulation to Restore Hand Function in Children with Spinal Cord Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Goutam Singh, Assistant Professor, University of Louisville
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 24.0267
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-07

CONDITIONS: Spinal Cord Injury Cervical
Keywords: Pediatric onset; Transcutaneous spinal cord stimulation; Hand and arm function; Chronic spinal cord injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Activity based upper extremity training (Active Comparator): Activity-based upper extremity training (AB-UET) will be administered 5d/week and 1 hour 30 minutes/session.
  Interventions: Device: Activity based upper extremity training with and without stimulation
- Activity based upper extremity training with stimulation (Experimental): Activity-based upper extremity training (AB-UET + scTS) will be administered 5d/week and 1 hour 30 minutes/session. UE tasks will be repeated with and without scTS so that scTS is administered intermittently for the duration of ~ 10 minute/bouts.
  Interventions: Device: Activity based upper extremity training with and without stimulation

INTERVENTIONS:
Device: Activity based upper extremity training with and without stimulation — Activity-based upper extremity training (AB-UET) will be administered 5d/week and 1 hour 30 minutes/session. For AB-UET+ stimulation (scTS), UE tasks will be repeated with and without scTS so that scTS is administered intermittently for the duration of ~ 10 minute/bouts.

SUMMARY:
The main goal of this pilot study is to find the best ways to use transcutaneous spinal cord stimulation (scTS) to improve hand function in children with spinal cord injuries (SCI). The investigators will start by exploring the best places and strengths for applying scTS on the neck, the added benefits of applying scTS on the lower back (T11-T12), and comparing the effects of using activity based upper extremity training (a control treatment) alone versus combining it with scTS to help children with chronic SCI regain hand function.

DETAILED DESCRIPTION:
After learning about the study and potential risks, parents/legal guardians and their eligible children with SCI will sign consent and assent forms, respectively. For the first two aims of the study, the investigators will recruit and enroll 10 participants. In the first week, participants will undergo clinical assessments from day 1 to day 4 to categorize the severity and level of their injuries and assess their current arm and hand function. On day 5, eligible participants will have experimental assessments to measure hand grip and control, both with and without spinal cord stimulation (scTS) at one or two neck sites optimized to improve hand grip. On day 6, participants will have similar assessments, this time adding stimulation to the trunk area to help with upright sitting and study its impact on hand grip and control.

For the third aim, 4 participants who showed improved hand grip and control with stimulation in aims 1 and 2 will be selected on a first-come, first-served basis. They will undergo 20 sessions of activity-based upper extremity training, followed by 20 more sessions with the optimal stimulation sites identified from aims 1 and 2. After completing the training, participants will be asked to follow up and repeat experimental and clinical assessments to determine how long the improvements last.

ELIGIBILITY:
Inclusion Criteria:

For aim 1 and 2, 10 participants with SCI:

1. age 7-12 years;
2. chronic (>6 months), acquired upper motor neuron SCI;
3. cervical SCI at or above C8 neurological level with motor score of 1-3 for finger flexors
4. Pediatric Neurorecovery scale score of ≥2B and ≤ 4C for impaired grip

For Aim 3, 4 participants with SCI who:

1. complete aim 1 and 2;
2. consent/assent for aim 3
3. demonstrate a minimum of 10% increase in HG force with scTS (aim1-2)
4. confirmed volitional activation in hand muscles during hang grip assessment without scTS

Exclusion Criteria:

For all 3 aims will include:

1. Botox use within past 3 months (for upper or lower extremity);
2. current oral baclofen (or pump);
3. musculoskeletal impairment limiting range of motion;
4. unhealed fracture or other medical condition limiting participation in AB-UET;
5. etiology of spina bifida;
6. total ventilator dependence.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Hand grip | 12 weeks
  Voluntary maximal hand grip force
Hand control | 12 weeks
  Peak to peak distance on hand grip force

SECONDARY OUTCOMES:
Functional neurophysiological assessment-Upper extremity | 12 weeks
  Multi-muscle activation patterns
Pediatric Neurorecovery scale | 12 weeks
  Pediatric Neurorecovery scale (NRS) is a validated clinical scale that assesses a child's (age 1-12 years) neuromuscular capacity to perform everyday tasks without behavioral compensation, physical assistance, or assistive device. The total score is the sum of all tasks on a scale from 1-12. For a total of 12 items, the highest score being 144 and lowest a sore of 12. Higher scores indicate improved function.
Capabilities of upper extremity test | 12 weeks
  The Capabilities of the Upper Extremity Test (CUE-T) is a performance measure intended to assess upper extremity function following spinal cord injury. The CUE-T is an objective measure of the ability to complete actions and tasks involving the arm and hand in individuals with tetraplegia and can be used clinically, for research and in clinical trials. Respondents answer questions on a 7-point scale that represents their self-perceived difficulty in performing the action, with 1 indicating "totally limited, can't do at all" and 7 indicating "not at all limited". The total score is the sum of all responses, and ranges from 32 to 224, with higher scores indicating greater function.
Box and block test | 12 weeks
  The Box and Block Test (BBT) measures unilateral gross manual dexterity and is validated in pediatric population. The score is the number of blocks carried from one compartment to the other in one minute. Each hand is scored separately. Higher scores within 1-minute indicate better manual dexterity.

CONTACTS AND LOCATIONS:
Overall Officials: Goutam Singh, PhD, Principal Investigator — University of Louisville and Spalding University